CLINICAL TRIAL: NCT05975983
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of INS018_055 Administered Orally to Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Study Evaluating INS018_055 Administered Orally to Subjects With Idiopathic Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: InSilico Medicine Hong Kong Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS018-055-004
Record Dates: First submitted 2023-07-27; First posted 2023-08-04 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis; Fibrosis; Pathologic Processes; Lung Diseases, Interstitial; Lung Diseases; Respiratory Tract Diseases
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis; Fibrosis; Pathologic Processes; Lung Diseases, Interstitial; Lung Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INS018_055 (Experimental): INS018_055 is administered once daily up to 12 weeks
  Interventions: Drug: INS018_055
- Placebo (Placebo Comparator): Placebo is administered once daily up to 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INS018_055 — Pharmaceutical formulation: Tablet
  Mode of Administration: Oral
  Arms: INS018_055
Drug: Placebo — Pharmaceutical formulation: Tablet
  Mode of Administration: Oral
  Arms: Placebo

SUMMARY:
The purpose of this revised Phase IIa study is to demonstrate safety of INS018_055 over 12 weeks in adults with Idiopathic Pulmonary Fibrosis (IPF).

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis is a fatal lung disease characterized by reduced quality of life (QoL) and a median survival of 3 to 4 years. While current standard of care (SoC) treatments including pirfenidone and nintedanib slow disease progression, they are not curative and poorly tolerated due to their toxicity profiles. To address the need for new treatments in IPF, InSilico Medicine is developing INS018_055, a potent inhibitor of the serine/threonine kinase Traf2- and Nckinteracting kinase (TNIK).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥40 years based on the date of the written informed consent form
2. Diagnosis of IPF as defined by American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association guidelines
3. In a stable condition and suitable for study participation based on the results of medical history, physical examination, vital signs, 12-lead ECG, and laboratory evaluation
4. Meeting all of the following criteria during the screening period:

   1. FVC ≥40% predicted normal
   2. DLCO corrected for Hgb ≥25% and <80% predicted normal
   3. Forced Expiratory Volume in the first second/FVC (FEV1/FVC) ratio >0.7 based on pre-bronchodilator value

Exclusion Criteria:

1. Acute IPF exacerbation within 4 months prior to Visit 1 and/or Day 1, as determined by the investigator
2. Patients who are unwilling to refrain from smoking within 3 months prior to screening and until the end of the study
3. Female patients who are pregnant or nursing
4. Abnormal ECG findings

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who have at least 1 treatment-emergent adverse event (TEAE) | Day 1 (Visit 2) up to Week 12 (End of Treatment (EOT))

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Time to reach maximum plasma concentration (Tmax) of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Area under the plasma concentration-time curve from time zero to dosing interval τ (AUC0-τ) of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Area under the plasma concentration-time curve from time zero to time with last measurable concentration t (AUC0-t) of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Area under the plasma concentration-time curve from time zero to infinity (∞) (AUC0-∞) of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Terminal elimination half-life (t1/2) of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Terminal elimination rate constant (λz) of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Apparent clearance (CL/F) of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Apparent volume of distribution (Vz/F) of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Accumulation ratio (Rac) for Cmax and AUC of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Trough plasma concentration (Ctrough) of INS018_055 and its major metabolites (INS018_063 and INS018_095) | Following the first dose on Day 1 (Visit 2) and the last dose during Week 12 (Visit 8, End of Treatment (EOT))
Relative change in Forced Vital Capacity (FVC) in mL | Week 0/Visit 2 up to Week 12
Percentage change in FVC in mL | Week 0/Visit 2 up to Week 12
Absolute and relative change in FVC % predicted | Week 0/Visit 2 up to Week 12
Change in Diffusion Capacity of the lung for Carbon Monoxide (DLCO) % predicted | Week 0/Visit 2 to Week 12
Change in Leicester Cough Questionnaire (LCQ) | Week 0 to Week 4, 8 and 12
Change in 6-Minute Walk Distance (6MWD) in meters | Week 0 to Week 12
Number of acute IPF exacerbations | Week 0 up to Week 12
Number of days hospitalized for acute IPF exacerbations | Week 0 to up Week 12

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Keck School of Medicine of USC, Los Angeles, California
  - Florida Lung Asthma and Sleep Specialist, Celebration, Florida
  - Central Florida Pulmonary Group, P.A. (CFPG) - Downtown Orlando, Orlando, Florida
  - Southeastern Research Center, Winston-Salem, North Carolina
  - University of Oklahoma Health Sciences Center (OUHSC), Oklahoma City, Oklahoma
  - Temple University Hospital-Temple Lung Center, Philadelphia, Pennsylvania
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Research Centers of America, McKinney, Texas

IPD SHARING:
Plan to Share IPD: No